CLINICAL TRIAL: NCT07275268
Title: DIAGNOSTIC CONTRIBUTION OF EARLY ABDOMINAL ULTRASOUND IN THE SITUATION OF ACUTE ABDOMEN OF PREMATURE
Acronym: EchoPrémA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2025/979
Record Dates: First submitted 2025-11-28; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-11

CONDITIONS: Acute Abdomen in Children

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Abdominal Ultrasound (Experimental): Abdominal Ultrasound
  Interventions: Procedure: Abdominal Ultrasound

INTERVENTIONS:
Procedure: Abdominal Ultrasound — Abdominal Ultrasound

SUMMARY:
This study will assess the diagnostic contribution of early abdominal ultrasound for acute abdomen in premature newborns.

Early ultrasound assessment would provide diagnostic assistance, in conjunction with clinical examination and biological testing, in the three main clinical situations encountered with an acute abdomen in premature infants: enterocolitis (digestive translocation of a bacterium secondary to inflammation, local fragility of the digestive tract, associated ischemic phenomena), reflex ileus (decrease in intestinal peristalsis secondary to peritoneal reactivity following inflammatory phenomena) and digestive immaturity (expressed by bloating, regurgitation, absence of spontaneous transit, related to the degree of prematurity).

ELIGIBILITY:
Inclusion Criteria:

Premature under 37 weeks of amenorrhea with an adverse event of special interest such as :

* altered abdomen with bloating or presence of previsouly unknow marked collateral circulation,
* absence of spontaneous transit (> 48 hours),
* episode of rectal bleeding,
* repeated regurgitation/vomiting (during more than 50% of feedings),
* prolonged fasting (>12 hours), OR
* increase in cardiorespiratory events on continuous monitoring associated with one of the elements listed above.

Exclusion Criteria:

* organic malformation detected during prenatal monitoring or discovered in the immediate postnatal period,
* chromosomal abnormality detected during prenatal monitoring or discovered in the immediate postnatal period,- spontaneous perforation occurring during the first week of life.

Max Age: 36 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Presence or absence of echographic signs | Day 5
  Presence of "positive" echographic signs such as:
  aeroportia, pneumatosis parietalis, pneumoperitoneum, bowel wall thickening, fluid effusion, distension of bowel loops, during the early echography for premature newborns with digestive symptomatology.

CONTACTS AND LOCATIONS:
Overall Officials: Chloé HILD, MD, Principal Investigator — CHU de Besançon; Marion AUBER LENOIR, MD, Principal Investigator — CHU de Besançon

IPD SHARING:
Plan to Share IPD: No